CLINICAL TRIAL: NCT02334215
Title: A Randomized Trial of Interim Methadone and Patient Navigation Initiated in Jail
Acronym: SOMATICS FRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Laura and John Arnold Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 3U01DA013636 (NIH); 3U01DA013636 (NIH)
Record Dates: First submitted 2014-09-26; First posted 2015-01-08 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methadone; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Methadone plus Patient Navigation (Experimental): Participants will begin methadone treatment during detention and will have a patient navigator for up to 3 months post-release from detention.
  Interventions: Drug: Methadone; Behavioral: Patient Navigation
- Methadone (Experimental): Participants will begin methadone during detention.
  Interventions: Drug: Methadone
- Enhanced Treatment as Usual (Active Comparator): Participants will receive opioid detoxification during detention, as well as drug abuse education, overdose prevention education, and referral to drug abuse treatment and overdose prevention services in the community.
  Interventions: Behavioral: Enhanced Treatment as Usual (ETAU)

INTERVENTIONS:
Drug: Methadone — Interim methadone treatment (methadone without routine counseling) will be provided in jail. Methadone treatment with counseling will be continued in the community.
  Arms: Methadone; Methadone plus Patient Navigation
Behavioral: Patient Navigation — A patient navigator will assist the participant for the first three months after release from jail to enter and remain in methadone treatment in the community.
  Arms: Methadone plus Patient Navigation
Behavioral: Enhanced Treatment as Usual (ETAU) — Participants will receive methadone detoxification, drug abuse and overdose prevention information, drug treatment and overdose prevention referral in the community.
  Arms: Enhanced Treatment as Usual

SUMMARY:
The purpose of this study is to determine which of three approaches started in jail is more effective in treating opioid use disorder: (1) methadone treatment without counseling (termed interim methadone) coupled with case management (termed patient navigation); (2) interim methadone without patient navigation; (3) or an enhanced treatment as usual including opioid detoxification, overdose prevention and drug treatment information and referral.

DETAILED DESCRIPTION:
This study is part of the NIDA "Studies of Medication for Addiction Treatment in Correctional Settings (SOMATICS)" U01 Collaborative. Our distinct NIH-funded study at Friends Research Institute has been aligned with two other jail-based opioid treatment studies conducted by researchers at New York University (NYU) and at University of California Los Angeles (UCLA). SOMATICS seeks to harmonize assessments and interventions across the three research centers (RCs) and the three independent studies in order to leverage power, sample size, and increase the generalizability of findings. Each of the RCs in the SOMATICS cooperative will conduct their own individual trial, sharing one study arm with another RC, and several core assessments across all sites. The SOMATICS collaborative will have a common Statistical Analysis Plan and Data and Safety Monitoring Plan (DSMP) including a single DSMB. The collaborative primary and secondary outcomes across all sites are listed below:

Collaborative Primary Outcome Measure:

1. DSM-5 Opioid Use Disorder Diagnosis during the 30 days prior to the 6 months post-release follow-up assessment: Measured by: modified World Mental Health Composite International Diagnostic Interview.

Collaborative Secondary Outcome Measures:

1. Illicit Opioid use: measured by urine drug testing results at 6 months post-release
2. Number of days incarcerated: Measured by self-report during the 6 months post-release.
3. HIV risk behavior: Measured by self-report (Drug Risk Assessment Battery [RAB] Needle Use score) at the 6-month post-release follow-up assessment.
4. Number of days of Opioids, Cocaine, Alcohol, Benzodiazepines, and/or IV Drug Use: Measured by Time Line Follow Back at 6 months post-release follow-up (TLFB; NYU, UCLA) and ASI (FRI).
5. Non-opioid drug use (Cocaine, Amphetamines, and Benzodiazepines): measured by urine drug testing at 6 months post-release
6. Number of days in any drug abuse treatment: Measured by self-report at 6 months post-release.
7. Number of arrests: Measured by self-report data collected at 6 months post-release.
8. Craving scores (for NYU and UCLA sites only): Measured by self-report craving scale at 6 months post-release.
9. Non-lethal overdose (Yes/No): Measured by self-report during the 6 months post-release.
10. Lethal overdose (Yes/No): Measured by public records data reviewed at 6 months post-release.
11. WHO Quality of Life-BREF (WHOQOL-BREF) score: Measured by self-report at 6 months post-release.
12. Analyses of above self-same outcomes at 12 months follow-up.
13. Once the primary trial is complete, the site in Baltimore will collect longer-term outcome data at a 24-month follow-up point through funding from the Arnold Foundation.

ELIGIBILITY:
Inclusion Criteria:

* 1) Meets Diagnostic and Statistical Manual -5 (DSM-5) criteria for opioid use disorder; (2) detained for at least 48 hours; (3) receiving opioid withdrawal treatment (as-usual) through the Detention Center's medical providers; (4) able and willing to provide informed consent in English; (5) detained for a charge that, if found guilty, will result in a sentence of less than 1 year; (6) plan to reside in Baltimore upon release; (7) 18 years of age and older.

Exclusion Criteria:

* (1) enrolled in methadone or buprenorphine treatment in the community at the time of arrest; (2) having a medical (liver failure, congestive heart failure) or psychiatric condition (e.g., suicidal ideation, psychosis) that would make participation unsafe in the judgment of the medical staff or the PI; (3) pregnancy; (4) allergy to methadone; and, (5) requiring treatment for alcohol or sedative hypnotic withdrawal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore City Detention Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Mitchell MM, Kelly SM, O'Grady KE, Jaffe JH, Mitchell SG, Schwartz RP. HIV-Risk Behavior Among Adults with Opioid Use Disorder During 12 Months Following Pre-trial Detention: Results from a Randomized Trial of Methadone Treatment. AIDS Behav. 2021 Apr;25(4):1247-1256. doi: 10.1007/s10461-020-03090-y. Epub 2020 Nov 16. PMID 33196937
- [Derived] Schwartz RP, Kelly SM, Mitchell SG, O'Grady KE, Duren T, Sharma A, Gryczynski J, Jaffe JH. Randomized trial of methadone treatment of arrestees: 24-month post-release outcomes. Drug Alcohol Depend. 2021 Jan 1;218:108392. doi: 10.1016/j.drugalcdep.2020.108392. Epub 2020 Nov 2. PMID 33187759
- [Derived] Mitchell MM, Gryczynski J, Mitchell SG, Kelly SM, O'Grady KE, Monico LB, Schwartz RP. A Latent Class Analysis of HIV Risk Factors Among Men and Women with Opioid Use Disorder in Pre-trial Detention. AIDS Behav. 2020 Jun;24(6):1776-1783. doi: 10.1007/s10461-019-02726-y. PMID 31748939
- [Derived] Schwartz RP, Kelly SM, Mitchell SG, Dunlap L, Zarkin GA, Sharma A, O'Grady KE, Jaffe JH. Interim methadone and patient navigation in jail: Rationale and design of a randomized clinical trial. Contemp Clin Trials. 2016 Jul;49:21-8. doi: 10.1016/j.cct.2016.06.002. Epub 2016 Jun 7. PMID 27282117

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Started | 75 | 74 | 76
Completed (Number of participants that had at least one urine test conducted) | 68 | 68 | 61
Not Completed | 7 | 6 | 15
Not completed — Death | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 4
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Not released from incarceration on time | 3 | 3 | 3
Not completed — Incarcerated | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual | Total
Number analyzed (Participants) | 75 | 74 | 76 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (10.0) | 37.3 (10.0) | 37.9 (11.1) | 38.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 15 | 44
  Male | 60 | 60 | 61 | 181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3 | 6
  Not Hispanic or Latino | 72 | 74 | 73 | 219
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 51 | 45 | 43 | 139
  White | 17 | 17 | 22 | 56
  More than one race | 6 | 12 | 9 | 27
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75 | 74 | 76 | 225

OUTCOME MEASURES:

1. Primary Outcome: Predicted Probability Derived From the Generalized Linear Mixed Model of Opioid Urine Test Positive Results Over Time
Description: Predicted probability derived from the generalized linear mixed model opioid positive urine tests (0= negative; 1- positive) for heroin, oxycodone, methadone, or buprenorphine -- excluding the latter two positives when they results from prescribed medications to treat opioid use disorder)
Time Frame: 1, 3, 6, and 12 months post-release from incarceration
Population: The number analyzed at the follow-up points differ due to missing data (e.g., lost to follow-up, incarcerated individuals who were not drug tested, people interviewed by phone because they no longer lived in the area).
Measure: Least Squares Mean (Standard Error); unit: Probability
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 68 | 68 | 61
Probability
  1 month post-release from incarceration: number analyzed (Participants) | 54 | 53 | 38
  1 month post-release from incarceration | 0.70 (0.08) | 0.72 (0.09) | 0.66 (0.09)
  3 months post-release from incarceration: number analyzed (Participants) | 50 | 43 | 38
  3 months post-release from incarceration | 0.59 (0.08) | 0.72 (0.09) | 0.73 (0.08)
  6 months post-release from incarceration: number analyzed (Participants) | 52 | 44 | 44
  6 months post-release from incarceration | 0.49 (0.09) | 0.63 (0.10) | 0.71 (0.08)
  12 months post-release from incarceration: number analyzed (Participants) | 53 | 46 | 42
  12 months post-release from incarceration | 0.46 (0.08) | 0.71 (0.09) | 0.59 (0.09)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Contrast of interest: Methadone plus Patient Navigation and Methadone arms compared to Enhanced Treatment as Usual; Test type: Superiority; p = .32, Generalized Linear Mixed Model Analysis
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs. Methadone; Test type: Superiority; p = .32, Generalized Linear Mixed Model Analysis

2. Primary Outcome: Predicted Probability Derived From the General Linear Mixed Model of Entry Into Treatment for Opioid Use Disorder on the Methadone Treatment Exposure Form
Description: Predicted probability derived from the general linear mixed model of self-reported entry into treatment for opioid use disorder following release from incarceration and being in treatment 30 days post-release (0= no entry in treatment; 1= entry in treatment).
Time Frame: 30 days post-release from incarceration
Measure: Least Squares Mean (Standard Error); unit: Probability
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 61 | 56 | 50
Probability | 0.65 (0.09) | 0.62 (0.10) | 0.225 (0.09)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Contrast of Interest: Methadone plus Patient Navigation and Methadone Conditions combined vs. Enhanced Treatment as Usual Conditions; Test type: Superiority; p = .001, Generalized Linear Mixed Model Analysis
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs. Enhanced Treatment as Usual; Test type: Superiority; p = .84, Generalized Linear Mixed Model Analysis

3. Secondary Outcome: Predicted Probability Derived From Generalized Linear Mixed Model of Meeting Opioid Use Disorder Criteria as Determined by the Modified Composite International Diagnostic Interview (CIDI)
Description: Predicted probability derived from the Generalized Linear Mixed Model of meeting the Data and Statistical Manual - 5 criteria for Opioid Use Disorder in response to modified CIDI interview (0= does not meet criteria; 1= meets criteria).
Time Frame: one month period prior to the 3, 6, and 12 month post-release from incarceration
Population: The number analyzed at the follow-up points differ due to missing data (e.g., lost to follow-up, people who were incarcerated during the 30 days prior to the interview).
Measure: Least Squares Mean (Standard Error); unit: Probability
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 67 | 68 | 68
Probability
  3 months post-release from incarceration: number analyzed (Participants) | 55 | 57 | 43
  3 months post-release from incarceration | 0.66 (0.09) | 0.70 (0.08) | 0.76 (0.08)
  6 months post-release from incarceration: number analyzed (Participants) | 53 | 51 | 57
  6 months post-release from incarceration | 0.51 (0.09) | 0.59 (0.09) | 0.77 (0.08)
  12 months post-release from incarceration: number analyzed (Participants) | 58 | 52 | 52
  12 months post-release from incarceration | 0.54 (0.09) | 0.77 (0.11) | 0.59 (0.09)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Contrast of interest: Methadone plus Patient Navigation and Methadone Conditions combined vs. Enhanced Treatment as Usual; Test type: Superiority; p = 0.11, Generalized Linear Mixed Model Analysis
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs. Methadone; Test type: Superiority; p = 0.55, Generalized Linear Mixed Model Analysis

4. Secondary Outcome: Number of Participants With Arrests
Description: Official data on participant arrests subsequent to release from index incarceration.
Time Frame: one year post-release from incarceration
Population: Data presented on the subset of those participants who were released from index incarceration during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 71 | 69 | 72
Participants | 32 | 39 | 36
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Test type: Superiority; p = 0.55, Regression, Logistic
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs Methadone; Test type: Superiority; p = 0.57, Regression, Logistic

5. Secondary Outcome: Drug Risk Score on the Risk Assessment Battery (RAB)
Description: Drug Risk Scale Score on the Risk Assessment Battery. The scale's range goes from 0 to 22. Higher score represents greater frequency of drug risk behaviors
Time Frame: Baseline and 6, and 12 months post-release from incarceration
Population: The number analyzed at the follow-up points differ due to missing data (e.g., lost to follow-up, people who were incarcerated during the 6 months prior to the interview).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 76
score on a scale
  Baseline | 2.30 (.57) | 2.43 (.62) | 3.11 (.76)
  6 month post-release from incarceration: number analyzed (Participants) | 62 | 60 | 60
  6 month post-release from incarceration | 1.52 (.52) | 1.81 (.65) | 2.16 (.73)
  12 month post-release: number analyzed (Participants) | 64 | 58 | 57
  12 month post-release | .50 (.25) | 1.35 (.59) | 1.03 (.44)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Contrast of interest: Methadone plus Patient Navigation and Methadone compared to Enhanced Treatment as Usual; Test type: Superiority; p = .997, Generalized Linear Mixed Model
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs Methadone; Test type: Superiority; p = 0.26, Generalized Linear Mixed Model Analysis

6. Secondary Outcome: Sex Risk Score on the Risk Assessment Battery (RAB)
Description: Sex Risk Score on the Risk Assessment Battery (RAB). Higher scores represents greater risk. The score ranges from 0 to 18.
Time Frame: Baseline and 6, and 12 months post-release from incarceration
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 76
score on a scale
  Baseline: number analyzed (Participants) | 75 | 74 | 75
  Baseline | 4.52 (.34) | 4.78 (.35) | 4.68 (.34)
  6 months post-release: number analyzed (Participants) | 62 | 60 | 60
  6 months post-release | 3.93 (.34) | 3.94 (.35) | 4.27 (.36)
  12 month post-release: number analyzed (Participants) | 64 | 58 | 56
  12 month post-release | 3.78 (.36) | 4.61 (.42) | 4.17 (.38)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Test type: Superiority — Contrast of interest: Methadone plus Patient Navigation and Methadone compared to Enhanced Treatment as Usual; p = .663, Generalized Linear Mixed Model
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs Methadone; Test type: Superiority; p = 0.33, Generalized Linear Mixed Model Analysis

7. Secondary Outcome: Physical Domain Score on the World Health Organization Quality of Life Scale (WHOQOL-BREF)
Description: The score on the Physical Domain Scale of the World Health Organization Quality of Life Scale-BREF (WHOQOL-BREF). The scales range is from 0 to 100. The higher score represents better quality of life.
Time Frame: 1, 3, 6, and 12 months post-incarceration
Population: The number analyzed at the follow-up points differ due to missing data (e.g., lost to follow-up, people who were incarcerated during the 4 weeks prior to the interview).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 76
score on a scale
  Baseline | 54.6 (2.8) | 58.3 (3.0) | 57.1 (2.8)
  1 months post-release from incarceration: number analyzed (Participants) | 60 | 55 | 45
  1 months post-release from incarceration | 62.8 (3.0) | 62.2 (3.4) | 68.7 (3.4)
  3 months post-release from incarceration: number analyzed (Participants) | 55 | 57 | 43
  3 months post-release from incarceration | 60.3 (3.1) | 60.1 (3.1) | 67.3 (3.2)
  6 months post-release from incarceration: number analyzed (Participants) | 53 | 51 | 56
  6 months post-release from incarceration | 68.6 (3.1) | 66.3 (3.2) | 61.2 (3.0)
  12 months post-release from incarceration: number analyzed (Participants) | 58 | 52 | 52
  12 months post-release from incarceration | 63.1 (3.0) | 63.8 (3.2) | 60.3 (3.0)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Contrast of interest: Methadone plus Patient Navigation and Methadone arms compared to Enhanced Treatment as Usual; Test type: Superiority; p = 0.007, Generalized Linear Mixed Model Analysis
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs. Methadone; Test type: Superiority; p = .76, Generalized Linear Mixed Model Analysis

8. Secondary Outcome: Psychological Domain Score on the World Health Organization Quality of Life Scale (WHOQOL-BREF)
Description: Scale score on the Psychological Domain on the World Health Organization Quality of Life Scale (WHOQOL-BREF) goes from 1 to 100. The higher score represents a better quality of life.
Time Frame: 1, 3, 6, and 12 months post-release from incarceration
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 76
score on a scale
  Baseline | 56.8 (2.8) | 56.9 (3.0) | 55.9 (3.0)
  1 month post-release from incarceration: number analyzed (Participants) | 59 | 55 | 45
  1 month post-release from incarceration | 65.5 (3.1) | 64.0 (3.5) | 66.7 (3.5)
  3 months post-release from incarceration: number analyzed (Participants) | 55 | 57 | 43
  3 months post-release from incarceration | 62.6 (3.4) | 61.2 (3.3) | 66.6 (3.4)
  6 months post-release from incarceration: number analyzed (Participants) | 53 | 51 | 56
  6 months post-release from incarceration | 64.9 (3.5) | 63.9 (3.6) | 64.8 (3.4)
  12 months post-release from incarceration: number analyzed (Participants) | 58 | 52 | 52
  12 months post-release from incarceration | 62.0 (3.2) | 61.8 (3.4) | 64.4 (3.3)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Contrast of interest: Methadone plus Patient Navigation vs. Enhanced Treatment as Usual; Test type: Superiority; p = 0.60, Generalized Linear Mixed Model Analysis
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs. Methadone; Test type: Superiority; p = 1.0, Generalized Linear Mixed Model Analysis

9. Secondary Outcome: Social Domain Score on the World Health Organization Quality of Life Scale (WHOQOL-BREF)
Description: Social domain scale score on the World Health Organization Quality of Life Scale (WHOQOL-BREF) goes from 1 to 100. The higher score represents a better quality of life.
Time Frame: 1, 3, 6, and 12 month post-release from incarceration
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 76
score on a scale
  Baseline: number analyzed (Participants) | 75 | 55 | 45
  Baseline | 56.9 (3.9) | 57.7 (4.0) | 51.3 (3.9)
  1 month post-release from incarceration: number analyzed (Participants) | 60 | 74 | 76
  1 month post-release from incarceration | 63.6 (3.9) | 57.5 (4.4) | 64.9 (4.4)
  3 months post-release from incarceration: number analyzed (Participants) | 55 | 57 | 43
  3 months post-release from incarceration | 60.9 (4.1) | 62.4 (4.0) | 66.4 (4.1)
  6 months post-release from incarceration: number analyzed (Participants) | 53 | 51 | 56
  6 months post-release from incarceration | 63.3 (3.8) | 63.3 (3.9) | 58.8 (3.7)
  12 months post-release from incarceration: number analyzed (Participants) | 58 | 52 | 52
  12 months post-release from incarceration | 56.6 (4.3) | 55.4 (4.5) | 59.1 (4.3)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Contrast of interest: Methadone plus Patient Navigation and Methadone vs. Enhanced Treatment as Usual; Test type: Superiority; p = .09, Generalized Linear Mixed Model Analysis
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs. Methadone; Test type: Superiority; p = .74, Generalized Linear Mixed Model Analysis

10. Secondary Outcome: Environmental Domain Score on the World Health Organization Quality of Life Scale (WHOQOL-BREF)
Description: Environmental domain score on the World Health Organization Quality of Life Scale (WHOQOL-BREF) goes from 1 to 100. A higher score represents a better quality of life.
Time Frame: 1, 3, 6, and 12 months post-release from incarceration
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 76
score on a scale
  Baseline | 48.0 (3.0) | 54.6 (3.1) | 54.9 (3.0)
  1 months post-release from incarceration: number analyzed (Participants) | 60 | 55 | 45
  1 months post-release from incarceration | 56.1 (2.9) | 63.6 (3.3) | 65.1 (3.3)
  3 months post-release from incarceration: number analyzed (Participants) | 55 | 57 | 43
  3 months post-release from incarceration | 51.9 (3.2) | 55.1 (3.2) | 63.7 (3.3)
  6 months post-release from incarceration: number analyzed (Participants) | 53 | 51 | 56
  6 months post-release from incarceration | 59.0 (3.3) | 60.6 (3.4) | 57.2 (3.2)
  12 months post-release from incarceration: number analyzed (Participants) | 58 | 52 | 52
  12 months post-release from incarceration | 54.8 (3.2) | 59.4 (3.4) | 59.3 (3.3)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Contrast of interest: Methadone plus Patient Navigation and Methadone vs. Enhanced Treatment as Usual; Test type: Superiority; p = .013, Generalized Linear Mixed Model Analysis
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs. Methadone; Test type: Superiority; p = .71, Generalized Linear Mixed Model Analysis

11. Secondary Outcome: Overall Quality of Life Score on the World Health Organization Quality of Life Scale (WHOQOL-BREF)
Description: Self report quality of life as reported by participants following release from their index incarceration on a scale from 1 to 5. A higher score is a better outcome.
Time Frame: 1, 3, 6, and 12 month post-release from incarceration
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 76
units on a scale
  Baseline | 2.7 (1.6) | 2.8 (.16) | 3.1 (.16)
  1 month post-release from incarceration: number analyzed (Participants) | 60 | 55 | 45
  1 month post-release from incarceration | 3.49 (.162) | 3.56 (.19) | 3.40 (.19)
  3 months post-release from incarceration: number analyzed (Participants) | 55 | 57 | 43
  3 months post-release from incarceration | 3.15 (.17) | 3.46 (.17) | 3.57 (.17)
  6 months post-release from incarceration: number analyzed (Participants) | 53 | 51 | 56
  6 months post-release from incarceration | 3.51 (.17) | 3.58 (.18) | 3.53 (.17)
  12 months post-release from incarceration: number analyzed (Participants) | 57 | 52 | 52
  12 months post-release from incarceration | 3.29 (.17) | 3.43 (.18) | 3.45 (.17)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Test type: Superiority — Contrast of interest: Methadone plus Patient Navigation and Methadone vs. Enhanced Treatment as Usual; p = .32, Generalized Linear Mixed Model Analysis
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs. Methadone; Test type: Superiority; p = 0.85, Generalized Linear Mixed Model Analysis

12. Secondary Outcome: Predicted Probability Derived From the Generalized Linear Mixed Model of Being Retained in Treatment for Opioid Use Disorder on the Methadone Treatment Exposure Form
Description: Predicted Probability derived from the Generalized Linear Mixed of self-reported enrolled in treatment for Opioid Use Disorder at the time of the follow-up interview (0=not enrolled; 1=enrolled).
Time Frame: 12 months post-release from incarceration
Population: Participants who had completed at least one follow-up interview.
Measure: Least Squares Mean (Standard Error); unit: Probability
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 69 | 70 | 70
Probability
  1 month post-release from incarceration: number analyzed (Participants) | 61 | 56 | 50
  1 month post-release from incarceration | .63 (.08) | .56 (.09) | .26 (.08)
  3 months post-release from incarceration: number analyzed (Participants) | 60 | 61 | 52
  3 months post-release from incarceration | .57 (.08) | .47 (.09) | .19 (.07)
  6 months post-release from incarceration: number analyzed (Participants) | 60 | 59 | 59
  6 months post-release from incarceration | .52 (.09) | .52 (.09) | .24 (.07)
  12 months post-release from incarceration: number analyzed (Participants) | 64 | 58 | 58
  12 months post-release from incarceration | .40 (.09) | .27 (.09) | .29 (.08)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Test type: Superiority — Contrast of interest: Methadone plus Patient Navigation and Methadone vs. Enhanced Treatment as Usual; p = .10, Generalized Linear Mixed Model Analysis
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs. Methadone; Test type: Superiority; p = .74, Generalized Linear Mixed Model Analysis

13. Secondary Outcome: Mean Number of Days of Criminal Activity in the Past 30 Days Reported by Participants on the Addiction Severity Index (ASI)
Description: Mean number of days reported by participants of their criminal activity during the 30 days preceding the Addiction Severity Index interviews
Time Frame: 1, 3, 6, and 12 months post-release from incarceration
Population: Participants who completed at least one follow-up interview following release from index incarceration
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 76
Days
  1 month post-release from incarceration: number analyzed (Participants) | 60 | 55 | 45
  1 month post-release from incarceration | 5.22 (1.29) | 8.18 (1.74) | 8.22 (2.15)
  3 months post-release from incarceration: number analyzed (Participants) | 55 | 57 | 43
  3 months post-release from incarceration | 9.79 (1.81) | 9.35 (1.66) | 10.59 (2.15)
  6 months post-release from incarceration: number analyzed (Participants) | 53 | 51 | 57
  6 months post-release from incarceration | 9.24 (1.88) | 9.74 (1.89) | 11.49 (1.99)
  12 months post-release from incarceration: number analyzed (Participants) | 58 | 52 | 52
  12 months post-release from incarceration | 6.88 (1.54) | 9.97 (1.88) | 10.18 (1.99)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Test type: Superiority — Contrast of interest: Methadone plus Patient Navigation and Methadone vs. Enhanced Treatment as Usual; p = .42, Generalized Linear Mixed Model Analysis
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs. Methadone; Test type: Superiority; p = 0.42, Generalized Linear Mixed Model Analysis

14. Secondary Outcome: Mean Number of Days of Illicit Opioid Use Reported by Participants in the Past 30 Days
Description: Mean number of participant self-reported days of heroin use in the 30 days preceding the interview on the Addiction Severity Index (ASI)
Time Frame: 1, 3, 6, and 12 months post-release from incarceration
Population: Participants who were interviewed at least once following release from index incarceration.
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 76
Days
  1 month post-release from incarceration: number analyzed (Participants) | 60 | 55 | 45
  1 month post-release from incarceration | 8.66 (1.32) | 12.07 (1.72) | 14.88 (2.12)
  3 months post-release from incarceration: number analyzed (Participants) | 55 | 57 | 43
  3 months post-release from incarceration | 13.46 (1.84) | 15.15 (1.84) | 16.18 (2.04)
  6 months post-release from incarceration: number analyzed (Participants) | 53 | 51 | 57
  6 months post-release from incarceration | 13.56 (1.83) | 14.02 (1.90) | 15.42 (1.90)
  12 months post-release from incarceration: number analyzed (Participants) | 58 | 52 | 52
  12 months post-release from incarceration | 12.35 (1.66) | 14.70 (1.82) | 15.35 (1.90)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Test type: Superiority — Contrast of interest: Methadone plus Patient Navigation and Methadone vs. Enhanced Treatment as Usual; p = .28, Generalized Linear Mixed Model Analysis
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs. Methadone; Test type: Superiority; p = 0.44, Generalized Linear Mixed Model Analysis

15. Secondary Outcome: Participant Self-reported Mean Number of Days of Cocaine Use in the Past 30 Days
Description: Participant self-reported mean number of days of cocaine use in the 30 days preceding the interview on the Addiction Severity Index (ASI)
Time Frame: 1, 3, 6, and 12 months post-release from incarceration
Population: Participants who were interviewed at least once following release from index incarceration
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 76
Days
  1 month post-release from incarceration: number analyzed (Participants) | 60 | 55 | 45
  1 month post-release from incarceration | 5.95 (1.29) | 9.05 (1.73) | 11.01 (2.10)
  3 months post-release from incarceration: number analyzed (Participants) | 55 | 57 | 43
  3 months post-release from incarceration | 8.83 (1.71) | 11.32 (1.93) | 11.94 (2.14)
  6 months post-release from incarceration: number analyzed (Participants) | 53 | 51 | 57
  6 months post-release from incarceration | 10.74 (1.86) | 13.57 (2.23) | 11.94 (2.14)
  12 months post-release from incarceration: number analyzed (Participants) | 58 | 52 | 52
  12 months post-release from incarceration | 9.60 (1.70) | 14.46 (2.19) | 12.63 (2.01)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Contrast of interest: Methadone plus Patient Navigation and Methadone combined vs. Enhanced Treatment as Usual; Test type: Superiority; p = .61, Generalized Linear Mixed Model Analysis
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs. Methadone; Test type: Superiority; p = 0.72, Generalized Linear Mixed Model Analysis

16. Secondary Outcome: Predicted Probability Derived From the Generalized Linear Mixed Model of Meeting Cocaine Use Disorder Criteria in the Past 30 Days
Description: Predicted Probability Derived from the Generalized Linear Mixed Model meeting Data and Statistical Manual - 5 criteria for Cocaine Use Disorder on the modified Composite International Diagnostic Interview (CIDI) (0=Does not meet criteria; 1=meets criteria).
Time Frame: 3, 6, and 12 months post-release from incarceration
Population: Participants who completed at least one interview following release from index incarceration
Measure: Least Squares Mean (Standard Error); unit: Probability
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 75 | 74 | 76
Probability
  3 months post-release from incarceration: number analyzed (Participants) | 55 | 57 | 43
  3 months post-release from incarceration | .20 (.08) | .32 (.011) | .32 (.12)
  6 months post-release from incarceration: number analyzed (Participants) | 53 | 51 | 57
  6 months post-release from incarceration | .22 (.10) | .35 (.12) | .36 (.14)
  12 months post-release from incarceration: number analyzed (Participants) | 58 | 52 | 52
  12 months post-release from incarceration | .32 (.15) | .40 (.20) | .30 (.14)
Statistical Analysis 1: Comparison: Methadone Plus Patient Navigation vs Methadone vs Enhanced Treatment as Usual; Test type: Superiority — Contrast of interest: Methadone plus Patient Navigation and Methadone vs. Enhanced Treatment as Usual; p = .71, Generalized Linear Mixed Model Analysis
Statistical Analysis 2: Comparison: Methadone Plus Patient Navigation vs Methadone; Contrast of interest: Methadone plus Patient Navigation vs. Methadone; Test type: Superiority; p = .86, Generalized Linear Mixed Model Analysis

17. Secondary Outcome: Days of Hospitalization (Health Care Utilization) on the Economic Form 90 (EF-90)
Description: Mean number of days hospitalized during the 12 months post-release from incarceration
Time Frame: 12 months post-release from incarceration
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 67 | 67 | 58
Days | 2.0 (5.8) | 3.4 (9.7) | 1.2 (3.1)

18. Secondary Outcome: Cost of Substance Abuse Services
Description: Cost in US Dollars of substance abuse services on the modified Substance Abuse Services Cost Analysis Program
Time Frame: 12 months post-release from incarceration
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
Number analyzed (Participants) | 68 | 68 | 61
US Dollars | 3052 (533) | 2377 (351) | 1884 (292)

ADVERSE EVENTS:
Time Frame: 12 months following release from index incarceration
Arm/Group | Methadone Plus Patient Navigation | Methadone | Enhanced Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 1/75 | 3/74 | 3/76
Serious Adverse Events (participants affected / at risk) | 11/75 | 20/74 | 16/76
Other Adverse Events (participants affected / at risk) | 3/75 | 12/74 | 12/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methadone Plus Patient Navigation (N=75) | Methadone (N=74) | Enhanced Treatment as Usual (N=76)
Hospitalization (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalization (Infections and infestations) | 2 (3) | 7 (10) | 4 (8)
Hospitalization (Injury, poisoning and procedural complications) | 2 (2) | 2 (10) | 8 (8)
Hospitalization (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalization (Psychiatric disorders) | 1 (1) | 4 (7) | 1 (1)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (5) | 0 (0)
Hospitalization (Nervous system disorders) | 2 (3) | 2 (2) | 0 (0)
Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hospitalization (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Hospitalization (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Hospitalization (Cardiac disorders) | 2 (4) | 0 (0) | 0 (0)
Hospitalization (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methadone Plus Patient Navigation (N=75) | Methadone (N=74) | Enhanced Treatment as Usual (N=76)
Non fatal overdose (Injury, poisoning and procedural complications) | 3 | 12 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT02334215/Prot_SAP_000.pdf